CLINICAL TRIAL: NCT06683430
Title: High Potassium Diet Rich in Spices and Herbs-Salt Substitution (HPSH-SS) for Blood Pressure Reduction in Older Adults: Protocol for Diet Concept and Randomized Controlled Trial
Brief Title: High Potassium Diet with Spices and Herbs As Salt Substitute for Lowering Blood Pressure in Older Adults: Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Responsible Party: Principal Investigator, Farapti Farapti, Lecturer, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35/EC/KEPK/FKUA/2023
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Older Adults Institutionalized in Residential Homes
Keywords: sodium; potassium; spices and herbs; blood pressure; hypertension; elderly; protocol study; gerontology; dietary; anti-hypertensive; oxidative stress
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group High Potassium, Low Sodium Diet (Active Comparator): Participants received a diet enriched with potassium (3500 mg K) and reduced sodium (1500 mg Na) for 14 days.
  Interventions: Dietary Supplement: High Potassium, Low Sodium Diet
- Control Group Standard Diet (Low Potassium) (Placebo Comparator): Participants received a standard diet with low potassium (1700 mg K) and high sodium (2000 mg Na) daily for 14 days.
  Interventions: Dietary Supplement: Standard Diet

INTERVENTIONS:
Dietary Supplement: High Potassium, Low Sodium Diet — Daily intake of 3500 mg K and 1500 mg Na for 14 days.
  Arms: Intervention Group High Potassium, Low Sodium Diet
Dietary Supplement: Standard Diet — Daily intake of 1700 mg K and 2000 mg Na for 14 days.
  Arms: Control Group Standard Diet (Low Potassium)

SUMMARY:
This clinical trial aims to evaluate the High Potassium Diet Rich in Spices and Herbs-Salt Substitution (HPSH-SS) for reducing blood pressure in older adults. The study has two phases: the first focuses on developing a high-potassium, low-sodium diet, while the second involves a 14-day randomized controlled trial. Participants are divided into two groups: the intervention group (IG) receives an 1800 kcal daily diet with 3500 mg potassium and 1500 mg sodium, while the control group (CG) receives a diet with 1500 mg potassium and 2000 mg sodium. Key outcomes include changes in blood pressure, serum potassium, aldosterone, nitric oxide, and oxidative stress markers. The results could provide new dietary strategies for managing blood pressure in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* older adults aged ≥60 years residing in the nursing
* active and not bedridden
* without infectious disease, taste disorders, or dementia
* have blood pressure measurements indicating a systolic blood pressure (SBP) ≥130 mmHg and/or diastolic blood pressure (DBP) ≥85 mmHg

Exclusion Criteria:

* individuals with impaired kidney function (creatinine serum levels >1.2 mmol/L)
* uncontrolled diabetes mellitus (fasting blood sugar >126 mg/dL)
* obesity (BMI ≥30 kg/m2 )
* active smokers
* have memory impairment and depressive conditions
* participants declining continued participation, requiring intensive hospital care, or experiencing persistent vomiting and diarrhea were excluded from the intervention.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Change in Blood Pressure (mmHg) | Baseline, Day 8, and Day 15
  Measurement of the change in systolic and diastolic blood pressure from baseline to Day 8 and Day 15 to evaluate the effect of the high-potassium, low-sodium diet intervention.

SECONDARY OUTCOMES:
Change in Urinary Potassium Levels (mmol) | Baseline, Day 15
  All participants were provided with written and verbal instructions on the correct procedure for 24-hour urine collection to measure Na and K levels. Nurses were also instructed to assist participants with this process. Participants were asked to ensure accurate 24-hour urine collection and report any missing or uncollected urine. The urine samples were then transported by researchers to an internationally certified ISO 9001 labor laboratory for analysis of Na and K levels using the ion-selective electrode (ISE) method, which specifically responds to anions and cations. Urinary K levels were categorized as low (< 25 mmol), normal (25-125 mmol), and high (> 125 mmol).
Change in Urinary Sodium Levels (mmol) | Baseline, Day 15
  All participants were provided with written and verbal instructions on the correct procedure for 24-hour urine collection to measure Na and K levels. Nurses were also instructed to assist participants with this process. Participants were asked to ensure accurate 24-hour urine collection and report any missing or uncollected urine. The urine samples were then transported by researchers to an internationally certified ISO 9001 labor laboratory for analysis of Na and K levels using the ion-selective electrode (ISE) method, which specifically responds to anions and cations. Urinary Na levels were categorized as low (< 100 mmol), normal (100-260 mmol), and high (> 260 mmol).
Change in Serum Potassium Levels (mmol/L) | Baseline, Day 15
  Evaluation of changes in serum potassium levels as a response to dietary intake adjustments in the intervention group versus the control group. Serum potassium levels were determined through plasma blood testing using the ion-selective electrode (ISE) method. The samples were then transported by researchers to an internationally certified ISO 9001 laboratory. Plasma potassium levels were classified as follows: hypokalemia (< 3.5 mmol/L), normal (3.5-5 mmol/L), and hyperkalemia (> 5 mmol/L)
Change in Plasma Nitric Oxide Levels (µmol/L) | Baseline, Day 15
  Measurement of plasma nitric oxide to assess vascular response to the dietary intervention.
Change in Plasma F2-Isoprostane Levels (pmol/L) | Baseline, Day 15
  Analysis of changes in plasma F2-isoprostane as an oxidative stress marker to monitor the potential antioxidative effects of the dietary intervention.
Change in Plasma Aldosterone Levels (pmol/L) | Baseline, Day 15
  Measurement of plasma aldosterone levels to assess any physiological changes associated with potassium and sodium intake adjustments.
Change in Urinary Na/K Levels (mmol/L) | Baseline, Day 15
  The concentrations of sodium and potassium in urine were measured and expressed in millimoles per liter (mmol/L). The Na/K ratio in urine was calculated by dividing the sodium concentration by the potassium concentration. This ratio was used to evaluate the electrolyte balance in the study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- government institutional setting in Surabaya, Indonesia, namely Griya Wreda Surabaya nursing home., Surabaya, Jawa Timur, Angola

IPD SHARING:
Plan to Share IPD: No